CLINICAL TRIAL: NCT03101124
Title: Serum Concentration of Tranexamic Acid After Topical Administration in Massive Weight Loss Skin Reducing Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Aleris Helse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 270778; 2016-004246-28 (EudraCT Number)
Record Dates: First submitted 2017-03-30; First posted 2017-04-04 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Surgical Wound; Bleeding
Keywords: Hemostasis, Surgical; Tranexamic Acid; Antifibrinolytic Agents; Administration, Cutaneous; Administration, Intravenous; Administration, Topical
MeSH Terms: conditions — Surgical Wound; Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: 12 participants will be included in each of 3 groups: wound moistening group (skin reduction surgery), wound bolus group (after skin reduction surgery), and (for comparison) a group getting usual intravenous tranexamic acid before orthopedic surgery. It is not possible to conduct a formal power calculation, as it is completely unknown which concentrations could be expected after topical use; however, these concentrations are expected to be considerably lower than after intravenous use. Consequently, it is expected that the AUC values in all subjects in the topical (skin reducing surgery) group are far lower than in all subjects in the intravenous (orthopaedic surgery) group. 12 subjects is therefor considered an appropriate number.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- abdominoplasty moistening (Experimental): Tranexamic Acid 25 mg/ml for wound surface moistening prior to wound closure
  Interventions: Drug: Tranexamic Acid 25 mg/ml for wound surface moistening
- abdominoplasty bolus (Experimental): Tranexamic Acid 5 mg/ml as bolus in wound cavity after wound closure
  Interventions: Drug: Tranexamic Acid 5 mg/ml as bolus in wound cavity
- preoperative intravenous administration (Active Comparator): Tranexamic Acid Injectable Solution administered before hip replacement surgery
  Interventions: Drug: Tranexamic Acid Injectable Solution

INTERVENTIONS:
Drug: Tranexamic Acid 25 mg/ml for wound surface moistening — Wound surface moistened with 20 ml of tranexamic acid 25 mg/ml (total dose 500 mg) prior to wound closure
  Other Names: Cyclokapron
  Arms: abdominoplasty moistening
Drug: Tranexamic Acid 5 mg/ml as bolus in wound cavity — 200 ml of tranexamic acid 5 mg/ml (total dose 1 g) as a bolus instilled into the wound cavity after wound closure, which will remain in the cavity until the activation of drains one hour later
  Other Names: Cyclokapron
  Arms: abdominoplasty bolus
Drug: Tranexamic Acid Injectable Solution — 1 g of tranexamic acid administered intravenously in accordance with prevailing routines directly prior to planned surgical procedure.
  Other Names: Cyclokapron
  Arms: preoperative intravenous administration

SUMMARY:
Tranexamic acid is a drug that prevents clotted blood from dissolving and hence reduces bleeding. It is routinely given intravenously in many surgical situations where there is a risk of major bleeding. Concerns regarding possible adverse effects from intravenous use prevents a more widespread use, even in smaller surgeries. Topical application - using the drug directly on the wound surface- may give a higher concentration at the site of bleeding but a lower concentration in the rest of the body, and hence a lower risk of adverse effects. Here it will be investigated to what extent a defined dose of the drug is absorbed systemically - into the blood stream - when it is applied topically. This will then be compared to the concentration in the blood stream when administered intravenously. Blood samples will be obtained at defined time intervals after administration from patients receiving topical and patients receiving intravenous administration of the same single dose of tranexamic acid. Will less of the drug enter the blood stream if it is applied directly to the wound?

ELIGIBILITY:
Inclusion Criteria:

* planned for major skin reduction surgery (abdominoplasty/panniculectomy) after massive weight loss, or
* planned for orthopaedic hip replacement surgery

Exclusion Criteria:

* pregnancy
* breastfeeding
* known allergy to tranexamic acid/Cyklokapron®
* ongoing or former thromboembolic event
* known kidney failure, as defined by estimated glomerular filtration rate (eGFR)<60 ml/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Serum concentration of tranexamic acid | 24 hours
  as described by the Area Under the (time-concentration) Curve (AUC) from 0 to infinity, alternatively from 0 to 240 minutes if drug levels after 24 hours do not allow for such extrapolation

SECONDARY OUTCOMES:
AUC from 0 to 240 min | 24 hours
  if AUC from 0 to infinity turns out to be the primary end point.
Maximum concentration (Cmax) | 24 hours
  Maximal level of serum tranexamic acid in measurements
Timepoint for maximum serum concentration (Tmax) | 24 hours
  Timepoint for serum tranexamic acid read from AUC
Elimination half-life | 24 hours
  Reading elimination half-life from AUC
Adverse events | four weeks
  Possible adverse reactions or other complaints observed or reported by the patient - telephone interview
Adverse events | 1 day
  Possible adverse reactions or complaints observed or reported on the first postoperative day - clinical observation

CONTACTS AND LOCATIONS:
Overall Officials: Birger Henning Endreseth, MD PhD, Study Director — St. Olavs University Hospital
Locations (1):
- St Olavs Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ausen K, Pleym H, Liu J, Hegstad S, Nordgard HB, Pavlovic I, Spigset O. Serum Concentrations and Pharmacokinetics of Tranexamic Acid after Two Means of Topical Administration in Massive Weight Loss Skin-Reducing Surgery. Plast Reconstr Surg. 2019 Jun;143(6):1169e-1178e. doi: 10.1097/PRS.0000000000005620. PMID 31136475